CLINICAL TRIAL: NCT04209179
Title: A Randomized, Double-Blind, Multiple Ascending Oral Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of PCO371 in Patients With Hypoparathyroidism
Brief Title: A Clinical Study Investigating the Safety, Tolerability, PK and PD of PCO371 in Patients With Hypoparathyroidism
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated on the basis of the currently uncertain risk-benefit balance for the patients, and the strategic position of the development program
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: PCO104UG
Record Dates: First submitted 2019-11-28; First posted 2019-12-24 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Hypoparathyroidism
MeSH Terms: conditions — Hypoparathyroidism | interventions — PCO371

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PCO371 Low Dose and Low administration frequency (Experimental): PCO371 low dose and low administration frequency by oral administration for the first period ( Fixed-Dose treatment period). PCO371 will be titrated in the following period (Dose Titration Treatment period).
  Interventions: Drug: PCO371
- PCO371 High Dose and Low administration frequency (Experimental): PCO371 high dose and low administration frequency by oral administration for the first period ( Fixed-Dose treatment period). PCO371 will be titrated in the following period (Dose Titration Treatment period).
  Interventions: Drug: PCO371
- PCO371 High Dose and High administration frequency (Experimental): PCO371 high dose and high administration frequency by oral administration for the first period ( Fixed-Dose treatment period). PCO371 will be titrated in the following period (Dose Titration Treatment period).
  Interventions: Drug: PCO371
- Placebo (Placebo Comparator): Placebo by oral administration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PCO371 — PCO371 capsule
  Arms: PCO371 High Dose and High administration frequency; PCO371 High Dose and Low administration frequency; PCO371 Low Dose and Low administration frequency
Drug: Placebo — Placebo capsule
  Arms: Placebo

SUMMARY:
This is a multi-center, placebo-controlled, randomized, double-blind, multiple-ascending dose study in patients with hypoparathyroidism.

The total duration of study medication treatment will be 13 weeks and includes a Fixed-Dose Treatment period and a Dose Titration Treatment period. The Fixed-Dose Treatment period consists of multiple daily dosing at a fixed dose level. Once patients have completed the Fixed-Dose Treatment period, patients will enter the Dose Titration Treatment period where PCO371 (or placebo), oral calcium and oral active vitamin D can each be titrated according to the patient's albumin-corrected serum calcium level.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent, to use the device for PRO and electronic diary and to comply with the requirements of the protocol.
2. Adult males or females ≥18 years of age
3. History of hypoparathyroidism for more than 1-year post initial diagnosis
4. PTH level is inappropriately low
5. Dose of thyroid replacement therapy must have been stable for ≥3 months prior to first dose if receiving thyroid replacement therapy
6. Receiving treatment with active vitamin D therapy (calcitriol ≥0.25 μg/day or alfacalcidol ≥0.5 μg/day)
7. Receiving Oral calcium treatment (≥1000 mg/day)
8. No significant changes in the diet from 4 weeks prior to Screening and for the duration of the study.
9. Fasting albumin-corrected serum calcium concentration between 8.0 and 9.0 mg/dL at 2 consecutive visits during the Run-In period, and no more than 25% change in daily doses of oral Ca and active vitamin D between the 2 consecutive visits during the Run-In period.
10. On Day 1, fasting albumin-corrected serum calcium level between 7.5 and 9.0 mg/dL
11. Serum magnesium level ≥ lower limit of normal and ≤ 1.2 x laboratory upper limit of normal
12. Serum 25[OH] vitamin D level within the laboratory normal range
13. Estimated glomerular filtration rate ≥ 45 mL/min/1.73 m2
14. Women of childbearing potential must have a negative highly sensitive urine or serum pregnancy test result
15. For women of childbearing potential: agreement to use a highly effective contraceptive method during the treatment period and for 28 days after the last dose of study drug. Hormonal contraceptive methods must be supplemented by a barrier method (preferably male condom) and agreement to refrain from egg donation during the treatment period and for 28 days after the last dose of study drug.
16. For men: agreement to remain abstinent or use contraceptive measures. Men must refrain from donating sperm during this same period.
17. Ability to comply with the study protocol, in the investigator's judgment.
18. For Canadian sites only: Ferritin, as assessed by the local laboratory at screening, must be ≥ the lower limit of normal (LLN).

Exclusion Criteria:

1. Pregnant or breastfeeding or intending to become pregnant during the study or within 28 days after the last dose of PCO371
2. Known or suspected history of hypoparathyroidism resulting from an activating mutation in the Ca-sensing receptor gene or impaired responsiveness to PTH (pseudohypoparathyroidism)
3. Clinically significant hypomagnesemia. Adequately treated hypomagnesemia is permitted
4. Any disease that might affect calcium metabolism or calcium-phosphate homeostasis other than hypoparathyroidism
5. History of a major bone fracture within 3 months prior to Screening
6. Any history of clinically significant bleeding disorder or clinically significant abnormal clotting times
7. History of thyroid cancer unless documented to be disease free for ≥1 year
8. History of any other cancer in the past 3 years from Screening with the exception of thyroid cancer , completely removed nonmelanoma skin cancer, basal cell skin carcinoma, and cancer in situ of the cervix
9. Dependence on monthly or more frequent parenteral calcium infusions to maintain calcium homeostasis
10. Disease processes that may adversely affect gastrointestinal absorption
11. Use of oral bisphosphonates within 6 months of Screening and/or intravenous bisphosphonate preparations within 12 months of Screening. Any use of zoledronic acid prior to Screening.
12. Use of other drugs known to influence calcium and bone metabolism such as calcitonin, fluoride tablets or cinacalcet hydrochloride within 4 weeks prior to Screening.
13. Patients who have taken inducers of CYP3A4, Pgp,or BCRP within 1 month before IMP administration or taken inhibitors of CYP3A4, P-gp, or BCRP within 2 weeks before IMP administration (or either 6 times the t1/2 of the drugs mentioned above, whichever is longer).
14. Use of loop or thiazide diuretics within 14 days prior to first dose of IMP
15. Use of anti-coagulants, anti-platelet medications, and aspirin within 2 weeks (or within 6 times the t1/2 of the drug mentioned above, whichever is longer) prior to IMP administration
16. Use of proton pump inhibitors or H2 blockers within 48 hours prior to the first dose of IMP and antacids within 4 hours prior to the first dose of IMP.
17. History of radiotherapy to the skeleton within 5 years
18. Presence of open epiphyses at the distal radius and ulna as well as carpals, metacarpals, phalanges, and pelvis
19. ALT, AST, or ALP > 2.5 × ULN at Screening
20. Patients with documented active HBV, active HCV infection or any other known active virus infection considered to be clinically relevant by the investigator.
21. Evidence of active alcohol, drug, or other substance abuse or addiction
22. History of a seizure that is unrelated to hypocalcemia within 6 months prior to Screening
23. Insulin dependent diabetes mellitus or poorly controlled Type II diabetes mellitus (defined as hemoglobin A1c [HbA1c] >8%)
24. Chronic/severe cardiac disease
25. Active gout or history of active gout within 6 months prior to first dose of study medication
26. History of clinically significant cognitive deficit that would, at the discretion of the investigator, interfere with a patient's ability to participate in the trial.
27. Any disease or condition that, in the opinion of the investigator, has a high probability of precluding the patient from completing the study or where the patient could not or would not appropriately comply with study requirements
28. Participation in any clinical trials or has taken any IMP (including placebo) either within 2 months or 5 times the t1/2 of the IMP, whichever is longer, prior to first dose of IMP for this study
29. Previous treatment with PTH-like drugs, including PTH(1-84), PTH(1-34) or other Nterminal fragments or analogs of PTH or PTH-related proteins within 2 months or 5 times the t1/2 of the treatment (whichever is longer) prior to Screening.
30. Patients with hypersensitivity to PCO371 or to any component of this drug product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent adverse events | 13 weeks
  Treatment-emergent adverse events (TEAEs) will be assessed including the number and rate of TEAEs.
Selected adverse events | 13 weeks
  Hypercalcemia and hypocalcemia will be assessed including the number and rate of these.
Clinically significant change in the safety parameters; vital signs | 13 weeks
  Abnormal change in vital signs.
Clinically significant change in the safety parameters; body weight | 13 weeks
  Abnormal change in body weight.
Clinically significant change in the safety parameters; physical examination findings | 13 weeks
  Abnormal change in physical examination findings.
Clinically significant change in the safety parameters; laboratory test value | 13 weeks
  Abnormal change in laboratory test value including hematology, biochemistry, coagulation, urinalysis.
Clinically significant change in the safety parameters; electrocardiogram results | 13 weeks
  Abnormal change in electrocardiogram results including PQ (PR), RR, QRS, QT, pulse, QTcB, QTcF and ECG abnormalities.

SECONDARY OUTCOMES:
Pharmacokinetic data of PCO371; Plasma concentrations of PCO371 | 13 weeks
  Plasma concentrations versus time data
Pharmacokinetic data of PCO371; AUC0-last | 13 weeks
  AUC0-last of PCO371
Pharmacokinetic data of PCO371; Cmax of PCO371 | 13 weeks
  Cmax of PCO371
Pharmacokinetic data of PCO371; Tmax of PCO371 | 13 weeks
  Tmax of PCO371
Pharmacokinetic data of PCO371; T1/2 of PCO371 | 13 weeks
  T1/2 of PCO371
Pharmacodynamic data in serum or plasma | 13 weeks
  Time profile of serum/plasma concentrations in albumin corrected total calcium (Ca), 25 hydroxy vitamin D, 1,25-dihydroxy vitamin D, phosphate, magnesium, and cAMP
Pharmacodynamic data in urine | 13 weeks
  Urinary excretion of Ca, phosphate, magnesium, protein, sodium, potassium, chloride, and cAMP (via 24-hour urine collection)
Pharmacodynamic data; nephrogenous cAMP concentration | 13 weeks
  Time profile of nephrogenous cAMP concentration
Pharmacodynamic data; bone turnover markers in serum or plasma | 13 weeks
  Time profile of serum/plasma concentrations in bone turnover markers (i.e. bone-specific alkaline phosphatase, type 1 pro-collagen amino-terminal peptide, C-terminal telopeptide of type 1 collagen, and osteocalcin)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor Chugai Pharmaceutical Co. Ltd, Study Director — clinical-trials@chugai-pharm.co.jp
Locations (11):
- United States (8):
  - The Lundquist Institute, Torrance, California
  - University of Chicago, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
- Canada (2):
  - Endocrinologie et néphrologie Centre de recherche du CHU de Québec, Québec, CAN
  - McMaster University Bone Research & Education Centre, Oakville, Ontario
- Semmelweis Egyetem, Általános Orvostudományi Kar, Belgyógyászati és Onkológiai Klinika, Budapest, HU, Hungary

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). For further details on Chugai's Data Sharing Policy and how to request access to related clinical study documents, see here (www.chugai-pharm.co.jp/english/profile/rd/ctds_request.html).